CLINICAL TRIAL: NCT03311802
Title: A Risk Scores for Predicting Prevalence of Diabetes in the LAO Population
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: risk scores predicting DM
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2016-07

CONDITIONS: Undiagnosed Diabetes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This was a cross-sectional investigation conducted from December 2015 to July 2017, in 15 selected rural villages of 2 districts of Vientiane municipality, Lao PDR. Target population was interested people, both men and women of age range between 30 to 70 years, living in the selected community. Someone diagnosed with diabetes and/or using any anti-diabetic drug was excluded.

The study protocol initiated with the interview on demographic and behavior information with each participant, followed by physical exam and blood pressure measurement.

Fasting glucose were measured.

DETAILED DESCRIPTION:
All participants were invited to meet with the researcher.

Demographic data comprises of age, gender, family history of diabetes including parents and sibling, female with history of having baby weighing more than 4 kg, gestational diabetes, and history or current of dyslipidemia (triglycerides >150 mg/dl, LDL-C ≥ 100 mg/dl, HDL-c < 35 mg/dl), and behavior data were smoking habit, physical inactivity (less than 150 min/week or 3 day/week) were collected by interview.

After that each participant was appointed for blood pressure measurement. Body mass index was computed from body weight (kg) divided by body height (m2) using the weight and height scale.

Waist Circumference was measured at the midpoint between the superior border of iliac crest and the lowest rib using measuring tape with the subject in the position of standing relax and in underclothes

Hip circumference is measured at the level of maximal gluteal protrusion

Blood pressure (BP) value was done with the participants, after 5 minutes relaxing, sitting up right with their upper arm positioned at heart level and measured by Omron blood pressure monitor.

Fasting Plasma Glucose was utilized to identify an individual who is normal, has either pre-diabetes or undiagnosed diabetes. Venous blood samples were collected 5 ml from antecubital vein into the test tube

ELIGIBILITY:
Inclusion Criteria:

* of age range between 30 to 70 years, living in the selected community.

Exclusion Criteria:

* diagnosed with diabetes and/or using any anti-diabetic drug

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: population living in the selected community nearby Vientiane city
Sampling Method: Non-Probability Sample
Enrollment: 1098 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
fasting plasma glucose | 06.00-09.00 am
  overnight fasting blood glucose

IPD SHARING:
Plan to Share IPD: No